CLINICAL TRIAL: NCT02385123
Title: Evaluation of Human Immune Responses to Influenza Virus Vaccination in Healthy Volunteers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to COVID-19 pandemic.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-0071; HHSN272201400004C
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2018-11

CONDITIONS: Influenza; Influenza Immunisation
Keywords: ex-vivo; Healthy Volunteers; Immune Response; Influenza; plasmablasts; Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seasonal Flu Vaccine/Healthy Adult Volunteers (Experimental): 0.5 ml of seasonal inactivated influenza vaccine (IIV) was administered intramuscularly (IM) on Day 0 of each study season, for this multi-year study. A total of 60 participants were enrolled in this study.
  Interventions: Biological: Influenza Virus Vaccine Inactivated

INTERVENTIONS:
Biological: Influenza Virus Vaccine Inactivated — A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season.

SUMMARY:
This was an open label, single arm, Phase IV study of longitudinal immunologic responses to influenza vaccine in healthy adult participants, with the aim of enrolling up to 70 participants. This study enrolled males and non-pregnant females, 18-49 years old, inclusive. The participants were screened at enrollment with a history and physical exam and laboratory testing to ensure they were healthy enough to participate. Total enrollment was 60 participants.

Qualifying participants were vaccinated with an FDA approved seasonal inactivated influenza vaccine (IIV) according to the package insert. The study enrolled a total 60 participants. The primary objective of the study was to characterize HA-specific plasmablasts and memory B cells after influenza vaccination.

Note: Due to the Coronavirus Disease 2019 (COVID-19) pandemic, all non-essential research was halted in mid-March 2020. New enrollments were placed on hold for this study. Follow-up visits were also halted, which impacted the timing of participants' subsequent follow-up visits. Five participants had their Day 180 visits halted due to the COVID-19 pandemic.

DETAILED DESCRIPTION:
This was an open label, single arm, Phase IV study of longitudinal immunologic responses to influenza vaccine in healthy adult participants. This study enrolled males and non-pregnant females, 18-49 years old. The primary objective of the study was to characterize hemagglutinin (HA)-specific plasmablasts and memory B cells after influenza vaccination. The secondary objective was to investigate the longevity of humoral immunity to influenza virus in humans. Total enrollment was 60 participants.

This was a multi-year study. Participant duration in this study was 180 days. Participants were screened at enrollment with a history and physical exam and laboratory testing to ensure they were healthy enough to participate. Qualifying participants were vaccinated with an FDA approved seasonal inactivated influenza vaccine (IIV) according to the package insert. Approximately 450 ml of blood was collected for the research assays during the course of the study. Specifically, 16 ml was be collected for screening; 48ml was collected at enrollment; 96ml was collected at visit Days 7 and 14; and 64 ml was collected at 28, 90, and 180 days post vaccination.

A total of 60 participants were enrolled over the course of the study. Participants who completed the study were given the option to re-enroll in subsequent years as long as they continued to meet all inclusion/exclusion criteria. Re-enrolling participants were re-consented, given new participants identifiers, and counted towards the enrollment number goal for each year of participation. Safety was assessed from the time of study enrollment through the last study visit, via monitoring of vital signs, and querying for change in health status.

Note: Due to the Coronavirus Disease 2019 (COVID-19) pandemic, all non-essential research was halted in mid-March 2020. New enrollments were placed on hold for this study. Follow-up visits were also halted, which impacted the timing of participants' subsequent follow-up visits. Five participants had their Day 180 visits halted due to the COVID-19 pandemic.

A request was submitted to the Emory University Institutional Review Board to extend the missed visit windows for the Day 180 visit for a maximum of up to 90 days, to ensure that ample time would be available to bring participants back for their missed visits. Enrollment for this study ended on September 30, 2020, before research activities could resume at Emory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 49 years of age, inclusive.
* Subjects capable of providing written informed consent prior to initiation of any study procedures. Subjects able to understand and comply with planned study procedures and be available for all study visits.
* Screening labs within normal limits per the local laboratory normal ranges or considered to be not clinically significant by the investigator. Normal laboratory ranges are as listed below:

  * Hematology:

    * Hemoglobin: Male- 12.9-16.1 gm/dL, Female- 11.4-14.4 gm/dL
    * White blood cells (WBC): Male- 4.2-9.2 upper limit (uL), Female- 4-10 upper limit (uL)
    * Platelet count: 150-400 upper limit (uL)
  * Chemistries:

    * Kidney function: Glomerular filtration rate (GFR) > / = 60 mL/min/1.73 m^2;
    * Liver enzymes: Albumin > / = 3.5 g/dL; alanine aminotransferase (ALT) <66 U/L; aspartate aminotransferase (AST) <62 U/L
* Subjects who have not received the seasonal influenza vaccine in the current flu season and are not suspected to have had an influenza infection in the current flu season.
* Female subjects of child bearing potential must have a negative urine pregnancy test at the screening visit, enrollment visit and all subsequent study visits longer than 14 days since the last pregnancy test.

Exclusion Criteria:

* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV). This information will be obtained verbally from the patient.
* If female, active pregnancy or breast-feeding or plans to become pregnant during study participation.
* Chronic medical conditions that cause immunodeficiency or that require medications which could alter immune function such as immunosuppressants and immunoenhancers.
* Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation. This includes any chronic medical disease or condition, defined as persisting 3 months (defined as 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study
* Have an acute illness, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination. An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
* Persons taking anticoagulants, long-term aspirin therapy, or long-term systemic steroids (greater than 3 months in the past 12 months and any within 30 days).
* Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine;
* Have a known latex allergy;
* Have a history of severe reactions following previous immunization with licensed influenza virus vaccines.
* Have a history of Guillain-Barre syndrome.
* Subjects who had or are suspected to have had an influenza infection in the current influenza season.
* Subjects who, at screening, have abnormal vital signs and/or physical exam, including a temperature > / = 38.0 C, Systolic blood pressure < / = 90 or > / = 160 mmHg, pulse < / = 60 or > 110 beats per minute, new rash, signs of infection.
* Subjects who have already received the seasonal influenza vaccine in the current influenza vaccination season.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh Mehta, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital - W. Dean Warren General Clinical Research Center (GCRC), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Centers for Disease Control and Prevention (CDC). Prevention and control of seasonal influenza with vaccines. Recommendations of the Advisory Committee on Immunization Practices--United States, 2013-2014. MMWR Recomm Rep. 2013 Sep 20;62(RR-07):1-43. PMID 24048214
- [Background] Kunzel W, Glathe H, Engelmann H, Van Hoecke C. Kinetics of humoral antibody response to trivalent inactivated split influenza vaccine in subjects previously vaccinated or vaccinated for the first time. Vaccine. 1996 Aug;14(12):1108-10. doi: 10.1016/0264-410x(96)00061-8. PMID 8911005
- [Background] Pica N, Palese P. Toward a universal influenza virus vaccine: prospects and challenges. Annu Rev Med. 2013;64:189-202. doi: 10.1146/annurev-med-120611-145115. PMID 23327522

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The following methods were used to recruit participants: traditional flyers posted throughout campus, word of mouth referrals, and social media posts. In addition, listserves, and campus newsletters were also leveraged to expand our participant reach.
Groups:
- Seasonal Flu Vaccine/Healthy Adult Volunteers: This was an open label single arm study. For the purposes of this study, reportable adverse events were limited to any occurrence or worsening of an undesirable or unintended sign, symptom or disease that is specifically associated with a study procedure that is not part of the normal standard of care for the participant.
  There were minimal risks associated with venipuncture for obtaining research related labs. Foreseeable adverse events associated with venipuncture were: mild, temporary discomfort at the venipuncture site, bruising, and phlebitis. Very rarely, subjects may experience "vaso-vagal syndrome" during phlebotomy. Vaso-vagal reactions may include diaphoresis, nausea, syncope and rarely loss of consciousness.
  Anticipated adverse events related to administration of the inactivated influenza vaccine included: localized erythema, induration, swelling, itching and/or pain at the injection site, mild fever, myalgia, headache and malaise following vaccination.
  Since immunization with flu vaccine annually is offered as standard of care to healthy adults to prevent influenza infection, these anticipated reactions to the vaccine were not considered reportable adverse events. There were no illnesses requiring hospitalization that were deemed related to vaccination.
  Any adverse event listed by the vaccine manufacturer as a contraindication to further doses of the vaccine would have been considered an adverse event for the study.
Period: Overall Study
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Started | 60
Completed | 45
Not Completed | 15
Not completed — 15 participants were unable to complete study. Research was halted due to Coronavirus Disease 2019. | 15

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were measured for all 60 participants. All participants in this study received 0.5 ml of seasonal inactivated influenza vaccine (IIV), administered intramuscularly (IM) on Day 0 of each study season.
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.5 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 31
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Seroconversion (Pre-vaccination Hemagglutination Inhibition (HI) Titer <1:10 and a Post-vaccination HI Titer >1:40 or a Pre-vaccination HI Titer >1:10 and a Minimum Four-fold Rise in Post-vaccination HI Antibody Titer)
Description: Hemagglutination inhibition titers were measured against reference influenza A/H1N1 and A/H3N2 strains, as well as influenza B Yamagata lineage influenza strains. Strains were matched to the composition of the vaccine received by each subject. For H1N1 and H3N2, hemagglutination was performed using receptor destroying enzyme (RDE)-treated plasma and turkey red blood cells following the World Health Organization (WHO) standard protocol. For influenza B, guinea pig red blood cells were used instead.
Time Frame: Day 28
Population: Of the 60 donors enrolled in this study, 45 donors were eligible to have their samples analyzed for this time-point outcome measure. Donors who did not provide a sample for this time-point due to missing this time-point visit were not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Seasonal Flu Vaccine/Healthy Adult Volunteers: 0.5 ml of seasonal inactivated influenza vaccine (IIV) was administered intramuscularly (IM) on Day 0 of each study season.
  Influenza Virus Vaccine Inactivated: A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season.
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 45
Participants
  H1N1 seroconversion | 28
  H3N2 seroconversion | 30
  Influenza B Yamagata lineage seroconversion | 32

2. Primary Outcome: Percentage of Subjects With Pre-vaccination Titer <1:40
Description: Hemagglutination inhibition titers were measured against reference influenza A/H1N1 and A/H3N2 strains, as well as influenza B Yamagata lineage influenza strains. Strains were matched to the composition of the vaccine received by each subject. For H1N1 and H3N2, hemagglutination was performed using RDE-treated plasma and turkey red blood cells following the WHO standard protocol. For influenza B, guinea pig red blood cells were used instead.
Time Frame: Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 45
Participants
  A/H1N1 HAI titer <1:40 on day 0 | 24
  A/H3N2 HAI titer <1:40 on day 0 | 25
  B Yamagata lineage HAI titer <1:40 on day 0 | 13
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other; A single group analysis was used to determine this outcome measure. These are basic science, hypothesis-generating studies with limited numbers of participants and no control group. The outcomes have no comparisons built into them - the outcomes are stating what the cell counts are, what the antibody titers are, what percentage of people seroconverted, etc. As such, we cannot report any p-values etc. for comparisons (e.g. with unvaccinated people)

3. Secondary Outcome: Endpoint Immunoglobulin G (IgG) Titers for Serum Antibody Responses Directed Against the Full Length A/H1N1 Hemagglutinin (HA) Protein
Description: ELISAs were performed using serial dilutions of plasma incubated on Maxisorp ELISA plates coated with 50 nanograms per well of H1N1 hemagglutinin protein from strain A/Michigan/45/2015. Plasma samples were drawn from donors who received the 2017-18 or 2018-19 influenza vaccine. Bound serum IgG was detected using 1:1000 diluted goat anti-human IgG-horseradish peroxidase (HRP) from Jackson Immunoresearch and plates were developed using o-phenylenediamine (OPD) substrate and developed for 7 minutes. The ELISA endpoint titer was defined as the reciprocal dilution of plasma that produced a background-subtracted optical density at 490 (OD490) value of 0.3, corresponding to 10% of maximum binding. Endpoint titers were determined by interpolation from the serial dilution curve results using Graphpad Prism software.
Time Frame: Day 0
Population: Of the 60 donors for this study, 25 donors received the 2017-18 or 2018-19 vaccine. 1 donor did not have plasma samples available for all timepoints and was excluded from ELISA analysis.
Measure: Geometric Mean (Inter-Quartile Range); unit: H1 HA ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
H1 HA ELISA endpoint reciprocal dilution | 11851 [4170 to 39548]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Endpoint IgG Titers for Serum Antibody Responses Directed Against the Full Length A/H1N1 Hemagglutinin (HA) Protein
Description: ELISAs were performed using serial dilutions of plasma incubated on Maxisorp ELISA plates coated with 50 nanograms per well of H1N1 hemagglutinin protein from strain A/Michigan/45/2015. Plasma samples were drawn from donors who received the 2017-18 or 2018-19 influenza vaccine. Bound serum IgG was detected using 1:1000 diluted goat anti-human IgG-HRP from Jackson Immunoresearch and plates were developed using OPD substrate and developed for 7 minutes. The ELISA endpoint titer was defined as the reciprocal dilution of plasma that produced a background-subtracted OD490 value of 0.3, corresponding to 10% of maximum binding. Endpoint titers were determined by interpolation from the serial dilution curve results using Graphpad Prism software.
Time Frame: Day 180
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: H1 HA ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
H1 HA ELISA endpoint reciprocal dilution | 48445 [30675 to 78013]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Endpoint IgG Titers for Serum Antibody Responses Directed Against the Full Length A/H1N1 Hemagglutinin (HA) Protein
Description: as for outcome 4
Time Frame: Day 28
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: H1 HA ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
H1 HA ELISA endpoint reciprocal dilution | 121284 [66218 to 190689]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; A single group analysis was used to determine this outcome measure. These are basic science, hypothesis-generating studies with limited numbers of participants and no control group. The outcomes have no comparisons built into them - the outcomes are stating what the cell counts are, what the antibody titers are, what percentage of people seroconverted, etc. As such, we cannot report any p-values etc. for comparisons (e.g. with unvaccinated people

6. Secondary Outcome: Endpoint IgG Titers for Serum Antibody Responses Directed Against the H1N1 Hemagglutinin (HA) Stem Region
Description: ELISAs were performed using serial dilutions of plasma incubated on Maxisorp ELISA plates coated with 50 nanograms per well of a chimeric HA protein containing the head domain from an H6 influenza virus and the stem domain from A/California/07/2009. Plasma samples were drawn from donors who received the 2017-18 or 2018-19 influenza vaccine. Bound serum IgG was detected using 1:1000 diluted goat anti-human IgG-HRP from Jackson Immunoresearch and plates were developed using OPD substrate and developed for 7 minutes. The ELISA endpoint titer was defined as the reciprocal dilution of plasma that produced a background-subtracted OD490 value of 0.3, corresponding to 10% of maximum binding. Endpoint titers were determined by interpolation from the serial dilution curve results using Graphpad Prism software.
Time Frame: Day 0
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: stem ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
stem ELISA endpoint reciprocal dilution | 11140 [7032 to 22360]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

7. Secondary Outcome: Endpoint IgG Titers for Serum Antibody Responses Directed Against the H1N1 Hemagglutinin (HA) Stem Region
Description: as for outcome 6
Time Frame: Day 180
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: stem ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
stem ELISA endpoint reciprocal dilution | 16694 [7818 to 32048]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

8. Secondary Outcome: Endpoint IgG Titers for Serum Antibody Responses Directed Against the H1N1 Hemagglutinin (HA) Stem Region.
Description: as for outcome 6
Time Frame: Day 28
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: stem ELISA endpoint reciprocal dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 24
stem ELISA endpoint reciprocal dilution | 29905 [18411 to 42782]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

9. Secondary Outcome: Expression of Human Influenza-specific Monoclonal Antibodies From Plasmablasts
Description: Monoclonal antibodies were cloned from sorted H1 hemagglutinin-binding cells expressing high levels of the CD38 protein (CD38hi) plasmablasts isolated from a single donor on day 7 post vaccination.
Time Frame: Day 7
Population: Influenza-specific monoclonal antibodies (mAbs) were cloned from Day 7 plasmablasts from a single donor.
Measure: Number; unit: number of mAbs cloned
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 1
number of mAbs cloned | 6
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; A single group analysis was used to determine this outcome measure; Test type: Other; [other analysis details as in outcome 2, analysis 1]

10. Secondary Outcome: Frequency of Hemagglutinin (HA) Head-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: Peripheral blood mononuclear cells from volunteers who received the 2017-18 or 2018-19 influenza vaccine were stimulated with R-848/interleukin (IL)-2 to induce polyclonal plasmablast differentiation. Total H1-specific memory B cells were detected using hemagglutinin protein from A/Michigan/45/2015 as an ELISPOT capture antigen and IgG detection. Frequencies were expressed as a percentage of the spots observed using total IgG capture antibody. Head specific memory B cell frequencies were calculated by subtracting the percentage of stem-specific IgG memory B cells from the percentage of total H1-specific cells.
Time Frame: Day 0
Population: Of the 60 donors enrolled in this study, 25 donors received the 2017-18 or 2018-19 influenza vaccine. Two did not have peripheral blood mononuclear cell (PBMC) samples available at all timepoints and were excluded from analysis.
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.039 [0.027 to 0.063]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

11. Secondary Outcome: Frequency of Hemagglutinin (HA) Head-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: Peripheral blood mononuclear cells from volunteers who received the 2017-18 or 2018-19 influenza vaccine were stimulated with R-848/IL-2 to induce polyclonal plasmablast differentiation. Total H1-specific memory B cells were detected using hemagglutinin protein from A/Michigan/45/2015 as an ELISPOT capture antigen and IgG detection. Frequencies were expressed as a percentage of the spots observed using total IgG capture antibody. Head specific memory B cell frequencies were calculated by subtracting the percentage of stem-specific IgG memory B cells from the percentage of total H1-specific cells.
Time Frame: Day 180
Population: Of the 60 donors enrolled in this study, 25 donors received the 2017-18 or 2018-19 influenza vaccine. 2 did not have PBMC samples available at all timepoints and were excluded from analysis.
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.17 [0.084 to 0.32]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

12. Secondary Outcome: Frequency of Hemagglutinin (HA) Head-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: as for outcome 11
Time Frame: Day 28
Population: as for outcome 11
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.63 [0.27 to 1.50]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

13. Secondary Outcome: Frequency of Hemagglutinin (HA) Stem-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: Peripheral blood mononuclear cells from volunteers who received the 2017-18 or 2018-19 influenza vaccine were stimulated with R-848/IL-2 to induce polyclonal plasmablast differentiation. Stem-specific memory B cells were detected using a chimeric hemagglutinin containing an H6 influenza head domain and the stem domain from A/California/07/2009 as an ELISPOT capture antigen. Frequencies were expressed as a percentage of the spots observed using total IgG capture antibody.
Time Frame: Day 0
Population: as for outcome 11
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.023 [0.0094 to 0.041]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

14. Secondary Outcome: Frequency of Hemagglutinin (HA) Stem-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: as for outcome 13
Time Frame: Day 180
Population: as for outcome 11
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.088 [0.056 to 0.13]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

15. Secondary Outcome: Frequency of Hemagglutinin (HA) Stem-specific IgG Secreting Memory B Cells Per Total IgG Secreting Cells
Description: as for outcome 13
Time Frame: Day 28
Population: as for outcome 11
Measure: Geometric Mean (Inter-Quartile Range); unit: % of IgG memory B cells
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 23
% of IgG memory B cells | 0.17 [0.091 to 0.29]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

16. Secondary Outcome: Function of Human Influenza-specific Monoclonal Antibodies Assessed by Virus Neutralization Assay
Description: Madin-Darby canine kidney (MDCK) cells in 96-well plates were infected in duplicate for 5 hours with H1N1 influenza virus (strain A/Michigan/45/2015) that had been pre-incubated for 15 minutes at 37 degrees with influenza monoclonal antibodies. Pre-incubations were performed using serial 2-fold dilutions of each monoclonal antibody, beginning at a concentration of 30 micrograms per milliliter. Virus was used at a dose sufficient to yield 5% infection in the absence of antibody. Infection was assessed after 5 hours in methanol-permeabilized cells by staining with an influenza nucleoprotein-specific mouse antibody (HB65), then phycoerythrin (PE)-conjugated anti-mouse IgG, followed by identification of PE-positive cells by flow cytometry. The 50% neutralizing titer reported is equivalent to the lowest monoclonal antibody concentration that resulted in a greater than or equal to 2-fold reduction in viral infection relative to the no-antibody control.
Time Frame: Day 7
Population: All six antibodies were isolated from a single donor.
Measure: Median (Inter-Quartile Range); unit: 50% neutralizing conc. (micrograms/ml)
Units Other Than Participants: monoclonal antibodies
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 1
Number analyzed (monoclonal antibodies) | 6
50% neutralizing conc. (micrograms/ml) | 0.94 [0.58 to 1.9]

17. Secondary Outcome: Function of Human Influenza-specific Monoclonal Antibodies Assessed by Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Influenza-specific mAbs were assessed for HA binding by ELISA using recombinant HA protein from H1N1 strain A/California/07/2009. 50 ng of HA were coated per well in Maxisorp ELISA plates and serial dilutions of mAb were added. The concentration of each mAb that gave 50% maximal binding (EC50) was determined.
Time Frame: Day 7
Population: All six mAbs were isolated from a single donor.
Measure: Geometric Mean (Inter-Quartile Range); unit: ELISA EC50 titer in micrograms per ml
Units Other Than Participants: monoclonal antibodies
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 1
Number analyzed (monoclonal antibodies) | 6
ELISA EC50 titer in micrograms per ml | 0.13 [.087 to .274]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; These are basic science, hypothesis-generating studies with limited numbers of participants and no control group. The outcomes have no comparisons built into them - the outcomes are stating what the cell counts are, what the antibody titers are, what percentage of people seroconverted, etc. As such, we cannot report any p-values etc. for comparisons (e.g. with unvaccinated people)

18. Secondary Outcome: Function of Human Influenza-specific Monoclonal Antibodies Assessed by Hemagglutination Inhibition (HAI) Assay
Description: The HAI titer for each antibody was determined using the World Health Organization (WHO) standard protocol using H1N1 strain A/Michigan/45/2015.
Time Frame: Day 7
Population: All six mAbs were isolated from a single donor.
Measure: Median (Inter-Quartile Range); unit: HAI titer (micrograms per millliliter)
Units Other Than Participants: monoclonal antibodies
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 1
Number analyzed (monoclonal antibodies) | 6
HAI titer (micrograms per millliliter) | 7.5 [5 to 10]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 17, analysis 1]

19. Secondary Outcome: Quadrivalent Influenza Vaccine Immunoglobulin Gamma-1 (IgG1) ELISA Endpoint Titer
Description: ELISA titers were measured against the matched seasonal quadrivalent inactivated influenza vaccine received by each subject using a secondary antibody specific for human IgG1. The endpoint ELISA titer was defined as the reciprocal dilution of plasma that gave an optical density (OD) reading of 0.2, which corresponded to ~3 standard deviations above the background OD for ELISA wells incubated without plasma.
Time Frame: Day 0
Population: Samples were taken from donors who enrolled in the 2016-17 through 2019-20 seasons.
Measure: Geometric Mean (Inter-Quartile Range); unit: Reciprocal endpoint plasma dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 33
Reciprocal endpoint plasma dilution | 1877 [1435 to 2489]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — Single group analysis; [other analysis details as in outcome 2, analysis 1]

20. Secondary Outcome: Quadrivalent Influenza Vaccine IgG1 ELISA Endpoint Titer
Description: as for outcome 19
Time Frame: Day 180
Population: Samples were taken from donors who enrolled in the 2016-17 through 2018-19 seasons. Due to the COronaVIrus Disease of 2019 (COVID-19) pandemic, no samples could be drawn for this day 180 timepoint in the 2019-2020 season.
Measure: Geometric Mean (Inter-Quartile Range); unit: Reciprocal endpoint plasma dilution
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 17
Reciprocal endpoint plasma dilution | 3026 [2453 to 3722]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

21. Secondary Outcome: Quadrivalent Influenza Vaccine IgG1 ELISA Endpoint Titer
Description: as for outcome 19
Time Frame: Day 28
Population: Samples were taken from donors who enrolled in the 2016-17 through 2019-20 seasons.
Measure: Geometric Mean (Inter-Quartile Range); unit: reciprocal endpoint titer
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 32
reciprocal endpoint titer | 3744 [3018 to 4356]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

22. Secondary Outcome: Plasmablast Responses Against Hemagglutinin (HA) Head Antigens Assessed by Direct ex Vivo Enzyme-linked Immunospot (ELISPOT)
Description: Plasmablasts (PB) were enumerated directly from frozen PBMC without stimulation. Total H1-specific cells were detected using hemagglutinin protein from A/Michigan/45/2015 as an ELISPOT capture antigen and IgG detection. Frequencies were expressed as the number of spots observed per million peripheral blood mononuclear cells. Head specific PB frequencies were calculated by subtracting the number of stem-specific PB per million peripheral blood mononuclear cells from the number of total H1-specific PB per million cells.
Time Frame: Day 7
Population: Plasmablast responses to H1 head and stem were analyzed using day 7 PBMC from a subset of 14 donors who had a strong vaccine response to H1 hemagglutinin as determined by ELISA.
Measure: Geometric Mean (Inter-Quartile Range); unit: Head-specific IgG PB per million PBMC
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 14
Head-specific IgG PB per million PBMC | 1096 [635 to 2060]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

23. Secondary Outcome: Plasmablast Responses Against Hemagglutinin (HA) Stem Antigens Assessed by Direct ex Vivo Enzyme-linked Immunospot (ELISPOT)
Description: Plasmablasts (PB) were enumerated directly from frozen PBMC without stimulation. Stem-specific cells were detected using a chimeric hemagglutinin containing an H6 influenza head domain and the stem domain from A/California/07/2009 as an ELISPOT capture antigen and IgG detection. Frequencies were expressed as the number of spots observed per million peripheral blood mononuclear cells.
Time Frame: Day 7
Population: as for outcome 22
Measure: Geometric Mean (Inter-Quartile Range); unit: Stem-specific IgG PB per million PBMC
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
Number analyzed (Participants) | 14
Stem-specific IgG PB per million PBMC | 47.6 [15.5 to 98.5]
Statistical Analysis 1: Comparison: Seasonal Flu Vaccine/Healthy Adult Volunteers; Test type: Other — A single group analysis was used to determine this outcome measure; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months Adverse event data were collected from Day 0 (enrollment) to Day 180 (the end of follow-up). Adverse event data were collected at each of the follow-up visits (Day 7, Day 14, Day 28, Day 90, and Day 180).
Description: At each of the follow-up visits (Day 7, Day 14, Day 28, Day 90, and Day 180), participants were asked about any adverse events that they might have experienced since their last visit. Clinical health assessments were conducted at every study visit, and included inquiry regarding any illness, any change in medication, and any overall health changes since the last study visit. Adverse event data was collected from enrollment until the end of follow-up at Day 180.
Arm/Group | Seasonal Flu Vaccine/Healthy Adult Volunteers
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 9/60
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seasonal Flu Vaccine/Healthy Adult Volunteers (N=60)
Sore throat (pharyngitis) (Infections and infestations) | 2 (2) — 2 patients reported a sore throat. At Day 90, one patient reported sore throat. Onset was 7/14/2015, end date was 7/16/2015. At Day 180, one patient reported sore throat. Onset was 3/10/2018, end date was 3/17/2018. Deemed unrelated and mild.
Ear pain (Ear and labyrinth disorders) | 1 (1) — Ear pain
Urinary tract infection (Infections and infestations) | 1 (1) — One patient reported a urinary tract infection at Day 90. Start date was 1/3/2018. Stop date was 1/9/2018. Mild, deemed unrelated. Treatment required.
Influenza (General disorders) | 3 (3) — Three participants reported flu/flu-like symptoms. Deemed as mild and unrelated.
Foot pain (General disorders) | 1 (1) — One patient reported a foot injury that was incurred while fishing. Start date was 5/30/2015. End date was 5/30/2015. Mild, deemed unrelated, treatment required. Reported at Day 14.
Bell's Palsy (Nervous system disorders) | 1 (1) — One patient reported Bell's Palsy. Onset was 1/10/2017, resolved on 1/16/2017. Deemed unrelated. Treatment required.

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, all non-essential research was halted at our site (mid-March 2020). New enrollments and follow-up visits were halted, impacting the timing of participants' subsequent follow-up visits. There were participants whose Day 180 visits (final visits) were impacted. We requested an expansion of the Day 180 visit window. Due to the ongoing pandemic, our site was unable to resume participant research activities for this study, which closed to accrual on 3/31/2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT02385123/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02385123/ICF_001.pdf